CLINICAL TRIAL: NCT04241159
Title: A Small-Scale Study to Explore the Safety and Feasibility of Allogeneic Young Plasma Infusion in Older Adults Experiencing Disability Across the Spectrum of Frailty Syndrome
Brief Title: Study to Explore the Safety and Feasibility of Allogeneic Young Plasma Infusion in Older Adults
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Protocol required revisions and application was withdrawn from the IRB.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00061606
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2019-11

CONDITIONS: Frailty Syndrome; Heart Failure
Keywords: Frailty; Aging; Heart failure; Plasma; Infusion
MeSH Terms: conditions — Frailty; Heart Failure

STUDY DESIGN:
Intervention Model Description: All eligible study participants will undergo once weekly PF24 infusion for 8 weeks in the WFBH Clinical Research Unit (CRU), and return for cognitive, physical, and biomarker testing 1 week and 5 weeks after receiving the last dose of PF24.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Geriatric participants with frailty (Experimental): Geriatric participants aged 65-80 who have a diagnosis of frailty (Fried Frailty score of 3 or greater).
  Experimental dosing will consist of once weekly administration of PF24 over a period of 8 consecutive weeks (8 total doses over 56 days).
  Interventions: Biological: Allogeneic Young Plasma
- Geriatric participants with HFpEF (Experimental): Geriatric participants aged 65-80 who have a diagnosis of HFpEF.
  Experimental dosing will consist of once weekly administration of PF24 over a period of 8 consecutive weeks (8 total doses over 56 days).
  Interventions: Biological: Allogeneic Young Plasma

INTERVENTIONS:
Biological: Allogeneic Young Plasma — The experimental dosing will consist of once weekly administration of PF24 over a period of 8 consecutive weeks (8 total doses over 56 days). 250 mL single units of PF24 will be obtained from the South Texas Blood Bank and processed by the WFBH Blood Bank.
  1 unit (250 mL) PF24, will be infused at 1 mL/kg/hr, once weekly for 8 consecutive weeks.
  Other Names: PF24

SUMMARY:
Evaluate the feasibility of administering plasma (PF24) acquired from donors of a young chronological age intravenously to older adults at WFBMC while also exploring its effects on age-related functional decline

DETAILED DESCRIPTION:
A Small-Scale Study to Explore the Safety and Feasibility of Allogeneic Young Plasma Infusion in Older Adults Experiencing Disability Across the Spectrum of Frailty Syndrome

Plasma (PF24) will be transfused into enrolled male and female geriatric patients aged 65-80 who have a diagnosis of frailty (Fried Frailty score of 3 or greater) or HFpEF. The experimental dosing will consist of once weekly administration of PF24 over a period of 8 consecutive weeks (8 total doses over 56 days). Primary and secondary endpoints will measure safety and feasibility of infusing PF24 in this study population. Tertiary endpoints will include measurement of the Fried Frailty score, various cognitive testing, measurement of VO2max, and blood biomarkers associated with aging. We will measure change from baseline 1 week after the 8th infusion of PF24. Test of durability will occur 5 weeks after the 8th infusion of plasma.

ELIGIBILITY:
Inclusion Criteria:

* English speaking elderly males and females, aged 65-80 years, referred by the Gerontology Department and the Cardiology Clinic of the Wake Forest Baptist Health Sticht Center for Aging.
* a score of 3 or greater (at least frail status) as demonstrated by the Fried Frailty criteria.

Exclusion Criteria:

* Unable or unwilling to give informed consent in either study group
* Current psychiatric disorder not currently under control or being adequately treated
* Current consumption of more than 14 alcoholic drinks per week
* Self-reported inability to walk across a small room
* Residence in a nursing home
* Previous MOCA score below 21
* Difficulty in communication with study personnel due to speech or hearing problems
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
* Elective surgery, planned prior to signing consent
* Severe osteoarthritis
* Rheumatoid arthritis
* Severe B/L hip, knee, or hand pain (>7/10 on pain scale)
* Cancer requiring treatment in the past three years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Pulmonary disease including VQ mismatch/diffusion limitation, diminished inspired O2, hypoventilation, pulmonary fibrosis, or sarcoidosis
* Current tobacco use (smoke/chew)
* Currently prescribed corticosteroids
* Patients taking nucleoside analogues (Zebularine, 5-azaC, Decitabine)
* Patients on non-nucleoside analogues (Procaine, procainamide, hydralazine)
* History of an inherited bleeding disorder or vitamin K deficiency
* Cardiovascular disease (excluding HFpEF), clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator or uncontrolled angina.
* Parkinson's disease or other serious neurological disorder
* MMS score < 18
* Renal disease (any stage, inappropriate for age; Cr Cl < 60)
* Hypoalbuminemia, with serum albumin level < 3.5 g/dL
* History of IgA deficiency
* History of hypersensitivity to frozen plasma (PF24) or to plasma-derived products including any plasma protein
* Active hepatitis or history of liver transplant
* Anemia or polycythemia: Male - Hgb level below 12 or above 17.5 g/dL and/or HCT of 41%-53%. Female: Hgb level below 10.0 or above 16.0 g/dL and/or HCT 36%-46%
* Current use of anti-coagulants
* History of DMI or DMII
* Peripheral vascular disease
* Brain aneurysm or intracranial hemorrhage within the past 6 months
* History of Hepatitis B, Hepatitis C, or HIV infection
* Other illness of such severity that life expectancy is considered to be less than 12 months
* Patients with initial VO2max that falls below expected value or that does not meet a minimum VO2max of 20 mL * kg * min (in order to demonstrate a more clinically meaningful increase)
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg)
* CVA, hip fracture, B/L hip or knee replacement, or spinal surgery in the past 6 months
* Serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm) on ECG
* Myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolism in the past 6 months
* Undergoing physical therapy or cardiopulmonary rehabilitation
* Currently enrolled in another randomized trial involving lifestyle or pharmaceutical interventions
* Currently on an anaerobic/aerobic exercise plan
* Inability or unwillingness to return for all transfusions/FU visits

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | Post 5 weeks after the last infusion of plasma
  The primary outcomes of this phase 0 study are built upon evaluating the outcome of safety with administering plasma (PF24) acquired from donors of a young chronological age intravenously to older adults at WFBMC, as evidenced by lack of any grade 4-5 adverse events and >/=50% grade 3-4 adverse events, as defined by NCI CTCAE v5.0. Grade 1-2 events will be recorded for statistical purposes.

SECONDARY OUTCOMES:
Study participant retention | Post 5 weeks after the last infusion of plasma
  Secondary outcomes include indicators of feasibility as assessed by measuring study participant retention >/= 80%
Study participants ability to complete the Fried Frailty Assessment | Study endpoint weeks 11 and 15
  Measurement of the Fried Frailty Score - The stages of frailty based on the Fried Frailty assessment criteria: a score of 0 means that a person is robust or not frail. Persons with a score of 1 or 2 are at intermediate risk for adverse outcomes or are considered to be pre-frail. A score of 3-5 indicates that someone is frail

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Johnson, D.O.., M.S., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Aging Well in the 21st Century: Strategic Directions for Research on Aging. [cited 2018 8/10/18]; Available from: https://www.nia.nih.gov/about/aging-well-21st-century-strategic-directions-research-aging.
- [Background] Olivieri F, Capri M, Bonafe M, Morsiani C, Jung HJ, Spazzafumo L, Vina J, Suh Y. Circulating miRNAs and miRNA shuttles as biomarkers: Perspective trajectories of healthy and unhealthy aging. Mech Ageing Dev. 2017 Jul;165(Pt B):162-170. doi: 10.1016/j.mad.2016.12.004. Epub 2016 Dec 13. PMID 27986629
- [Background] Hayflick L. Biological aging is no longer an unsolved problem. Ann N Y Acad Sci. 2007 Apr;1100:1-13. doi: 10.1196/annals.1395.001. PMID 17460161
- [Background] Bilder, G., Human biological aging : from macromolecules to organ-systems. 2016, Hoboken, New Jersey: Wiley Blackwell. ix, 330 pages.
- [Background] Hatse S, Brouwers B, Dalmasso B, Laenen A, Kenis C, Schoffski P, Wildiers H. Circulating MicroRNAs as easy-to-measure aging biomarkers in older breast cancer patients: correlation with chronological age but not with fitness/frailty status. PLoS One. 2014 Oct 21;9(10):e110644. doi: 10.1371/journal.pone.0110644. eCollection 2014. PMID 25333486
- [Background] Kadota T, Fujita Y, Yoshioka Y, Araya J, Kuwano K, Ochiya T. Emerging role of extracellular vesicles as a senescence-associated secretory phenotype: Insights into the pathophysiology of lung diseases. Mol Aspects Med. 2018 Apr;60:92-103. doi: 10.1016/j.mam.2017.11.005. Epub 2017 Nov 20. PMID 29146100
- [Background] Sinha M, Jang YC, Oh J, Khong D, Wu EY, Manohar R, Miller C, Regalado SG, Loffredo FS, Pancoast JR, Hirshman MF, Lebowitz J, Shadrach JL, Cerletti M, Kim MJ, Serwold T, Goodyear LJ, Rosner B, Lee RT, Wagers AJ. Restoring systemic GDF11 levels reverses age-related dysfunction in mouse skeletal muscle. Science. 2014 May 9;344(6184):649-52. doi: 10.1126/science.1251152. Epub 2014 May 5. PMID 24797481
- [Background] Loffredo FS, Steinhauser ML, Jay SM, Gannon J, Pancoast JR, Yalamanchi P, Sinha M, Dall'Osso C, Khong D, Shadrach JL, Miller CM, Singer BS, Stewart A, Psychogios N, Gerszten RE, Hartigan AJ, Kim MJ, Serwold T, Wagers AJ, Lee RT. Growth differentiation factor 11 is a circulating factor that reverses age-related cardiac hypertrophy. Cell. 2013 May 9;153(4):828-39. doi: 10.1016/j.cell.2013.04.015. PMID 23663781
- [Background] Middeldorp J, Lehallier B, Villeda SA, Miedema SS, Evans E, Czirr E, Zhang H, Luo J, Stan T, Mosher KI, Masliah E, Wyss-Coray T. Preclinical Assessment of Young Blood Plasma for Alzheimer Disease. JAMA Neurol. 2016 Nov 1;73(11):1325-1333. doi: 10.1001/jamaneurol.2016.3185. PMID 27598869
- [Background] Katsimpardi L, Litterman NK, Schein PA, Miller CM, Loffredo FS, Wojtkiewicz GR, Chen JW, Lee RT, Wagers AJ, Rubin LL. Vascular and neurogenic rejuvenation of the aging mouse brain by young systemic factors. Science. 2014 May 9;344(6184):630-4. doi: 10.1126/science.1251141. Epub 2014 May 5. PMID 24797482
- [Background] Upadhya B, Pisani B, Kitzman DW. Evolution of a Geriatric Syndrome: Pathophysiology and Treatment of Heart Failure with Preserved Ejection Fraction. J Am Geriatr Soc. 2017 Nov;65(11):2431-2440. doi: 10.1111/jgs.15141. PMID 29124734
- [Background] Haykowsky MJ, Nicklas BJ, Brubaker PH, Hundley WG, Brinkley TE, Upadhya B, Becton JT, Nelson MD, Chen H, Kitzman DW. Regional Adipose Distribution and its Relationship to Exercise Intolerance in Older Obese Patients Who Have Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2018 Aug;6(8):640-649. doi: 10.1016/j.jchf.2018.06.002. Epub 2018 Jul 11. PMID 30007558
- [Background] Kitzman DW, Little WC, Brubaker PH, Anderson RT, Hundley WG, Marburger CT, Brosnihan B, Morgan TM, Stewart KP. Pathophysiological characterization of isolated diastolic heart failure in comparison to systolic heart failure. JAMA. 2002 Nov 6;288(17):2144-50. doi: 10.1001/jama.288.17.2144. PMID 12413374
- [Background] Haykowsky MJ, Tomczak CR, Scott JM, Paterson DI, Kitzman DW. Determinants of exercise intolerance in patients with heart failure and reduced or preserved ejection fraction. J Appl Physiol (1985). 2015 Sep 15;119(6):739-44. doi: 10.1152/japplphysiol.00049.2015. Epub 2015 Apr 24. PMID 25911681
- [Background] Stehle JR Jr, Leng X, Kitzman DW, Nicklas BJ, Kritchevsky SB, High KP. Lipopolysaccharide-binding protein, a surrogate marker of microbial translocation, is associated with physical function in healthy older adults. J Gerontol A Biol Sci Med Sci. 2012 Nov;67(11):1212-8. doi: 10.1093/gerona/gls178. Epub 2012 Sep 7. PMID 22960476
- [Background] Shah SJ, Kitzman DW, Borlaug BA, van Heerebeek L, Zile MR, Kass DA, Paulus WJ. Phenotype-Specific Treatment of Heart Failure With Preserved Ejection Fraction: A Multiorgan Roadmap. Circulation. 2016 Jul 5;134(1):73-90. doi: 10.1161/CIRCULATIONAHA.116.021884. PMID 27358439
- [Background] Kitzman DW, Upadhya B, Reeves G. Hospitalizations and Prognosis in Elderly Patients With Heart Failure and Preserved Ejection Fraction: Time to Treat the Whole Patient. JACC Heart Fail. 2015 Jun;3(6):442-444. doi: 10.1016/j.jchf.2015.01.009. Epub 2015 May 14. No abstract available. PMID 25982112
- [Background] Kitzman DW, Brubaker PH, Morgan TM, Stewart KP, Little WC. Exercise training in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. Circ Heart Fail. 2010 Nov;3(6):659-67. doi: 10.1161/CIRCHEARTFAILURE.110.958785. Epub 2010 Sep 17. PMID 20852060
- [Background] Kitzman DW, Brubaker P, Morgan T, Haykowsky M, Hundley G, Kraus WE, Eggebeen J, Nicklas BJ. Effect of Caloric Restriction or Aerobic Exercise Training on Peak Oxygen Consumption and Quality of Life in Obese Older Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Jan 5;315(1):36-46. doi: 10.1001/jama.2015.17346. PMID 26746456
- [Background] Triposkiadis F, Xanthopoulos A, Butler J. Cardiovascular Aging and Heart Failure: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Aug 13;74(6):804-813. doi: 10.1016/j.jacc.2019.06.053. PMID 31395131
- [Background] Justice JN, Ferrucci L, Newman AB, Aroda VR, Bahnson JL, Divers J, Espeland MA, Marcovina S, Pollak MN, Kritchevsky SB, Barzilai N, Kuchel GA. A framework for selection of blood-based biomarkers for geroscience-guided clinical trials: report from the TAME Biomarkers Workgroup. Geroscience. 2018 Dec;40(5-6):419-436. doi: 10.1007/s11357-018-0042-y. Epub 2018 Aug 27. PMID 30151729
- [Background] Savarese, D. Common Terminology Criteria for Adverse Events. 2019 [cited 2019 2019]; Available from: https://www.uptodate.com/contents/common-terminology-criteria-for-adverse-events?search=Common%20Terminology%20Criteria%20for%20Adverse%20Events.&source=search_result&selectedTitle=1~38&usage_type=default&display_rank=1
- [Background] Nicklas BJ, Wang X, You T, Lyles MF, Demons J, Easter L, Berry MJ, Lenchik L, Carr JJ. Effect of exercise intensity on abdominal fat loss during calorie restriction in overweight and obese postmenopausal women: a randomized, controlled trial. Am J Clin Nutr. 2009 Apr;89(4):1043-52. doi: 10.3945/ajcn.2008.26938. Epub 2009 Feb 11. PMID 19211823
- [Background] Misquita NA, Davis DC, Dobrovolny CL, Ryan AS, Dennis KE, Nicklas BJ. Applicability of maximal oxygen consumption criteria in obese, postmenopausal women. J Womens Health Gend Based Med. 2001 Nov;10(9):879-85. doi: 10.1089/152460901753285787. PMID 11747683
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Hobart MP, Goldberg R, Bartko JJ, Gold JM. Repeatable battery for the assessment of neuropsychological status as a screening test in schizophrenia, II: convergent/discriminant validity and diagnostic group comparisons. Am J Psychiatry. 1999 Dec;156(12):1951-7. doi: 10.1176/ajp.156.12.1951. PMID 10588410
- [Background] Silvergleid, A.J. Clinical Use of Plasma Components. [cited 2019]/ Available from: https://www.uptodate.com/contents/clinical-use-of-plasma-components
- [Background] The PLasma for Alzheimer SymptoM Amelioration (PLASMA) Study (PLASMA). Available from: https://clinicaltrials.gov/ct2/show/NCT02256306?term=PLASMA&rank=1
- [Background] Reversing Epigenetic & Other Markers of Senescence by Transfusing Young Plasma To Older Human Subjects (RESET-YOUTH). Available from: https://clinicaltrials.gov/ct2/show/NCT03353597?term=Reset-YOuth&rank=1
- [Background] Fresh frozen plasma: indications and risks. National Institutes of Health Consensus Development Conference Statement. Natl Inst Health Consens Dev Conf Consens Statement. 1984;5(5):4 p.. No abstract available. PMID 6395009
- [Background] Silvergleid, A.J. Approach to the patient with a suspected acute transfusion reaction. 4/23/18]; Available from: https://www.uptodate.com/contents/approach-to-the-patient-with-a-suspected-acute-transfusion-reaction
- [Background] Diane, S. Common Terminology Criteria for Adverse Events. April 23, 2018; Available from: http://www.uptodate.com